CLINICAL TRIAL: NCT05580094
Title: Combined General Anesthesia and Ultrasound Guided Supraclavicular Block Versus General Anesthesia in Pediatric Patients With Chronic Kidney Disease Undergoing Upper Limb Superficialization of Arteriovenous Fistula.
Brief Title: Combined Supraclavicular Block and General Anesthesia in Pediatric Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Fathy Radwan Abd Elzaher, Resident doctor at anesthesia,icu and pain management department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: supraclavicular block and GA
Record Dates: First submitted 2022-10-06; First posted 2022-10-14 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia only. (Placebo Comparator): the pediatric patients will receive general anesthesia only.
  Interventions: Other: general anesthesia only.
- General anesthesia plus supraclavicular block. (Active Comparator): the pediatric patients will receive combined supraclavicular block and general anesthesia.
  Interventions: Other: general anesthesia plus supraclavicular block.

INTERVENTIONS:
Other: general anesthesia only. — induction of general anesthesia by propofol and maintenance sevoflurane.
  Arms: General anesthesia only.
Other: general anesthesia plus supraclavicular block. — induction of general anesthesia by propofol and maintenance sevoflurane then the patients will receive the supraclavicular block with bupivacaine 0.5 ml per kg.
  Arms: General anesthesia plus supraclavicular block.

SUMMARY:
* compare the safety and efficacy of ultrasound-guided supraclavicular block in addition to general anesthesia in pediatric patients undergoing upper limb superficialization of arteriovenous fistula for hemodialysis.
* compare the amount of analgesic consumption as well as vasodilatation of upper limb blood vessels and its implications on the vascular anastomosis.

DETAILED DESCRIPTION:
Established renal disease is a signiﬁcant cause of morbidity and mortality in children and has implications for the conduct of general anesthesia (1).

Anesthetic management of pediatric patients is uniquely challenging. A large part of the anesthetic care includes pain management, management of concomitant disease, and risk reduction for adverse events. Perioperative pain management usually involves a multimodal pharmacologic approach to minimize opioid requirements. Regional anesthesia is valuable for postoperative pain control (2).

Postoperative analgesia is dictated by the extent and nature of the surgery. Regional block should be utilized where possible for its opioid-sparing effects. Where morphine infusions are commenced, the dose should be reduced due to the risk of accumulation of active metabolites and resultant opiate toxicity. Non-steroidal anti-inﬂammatory drugs are always avoided due to their deleterious effects on urine output (3).

Pediatric regional anesthesia is one of the most valuable and safe tools to treat perioperative pain and is an essential part of modern anesthetic practice. It provides excellent pain relief and allows caregivers to use multimodal analgesic techniques and decrease the use of opioids. Upper extremity brachial plexus blocks in children Various approaches to brachial plexus are available. The choice of the block is made depending on the indications. The supra-clavicular approach covers all the surgeries of the humerus and below (4).

The use of regional anaesthesia is mostly associated with vasodilatation which may guard against arterial spasm and may play a role in decreasing the postoperative complication and success of the superficialization of the arteriovenous shunt as a line for hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients of less than 18 years old.
* with chronic kidney disease.
* undergoing upper limb superficialization of arteriovenous fistula for haemodialysis.

Exclusion Criteria:

* Patient known to have allergy to the studied drugs.
* Patients with contraindications to regional anesthesia.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
brachiocephalic fistula maturation time | 6 month postoperative
  time in weeks required by fistula to be clinically mature

SECONDARY OUTCOMES:
anaesthetic consumption | 90 minutes intraoperative
  measurment of anesthesia MAC
postoperative analgesia time | 24 hours postoperative
EMERGENCE agitation | 30 minutes postoperative
  RASS score used with -5 = deeply sedated and 4 = highly agitated
VAS score | 24h postoperative
  scale of 10 points. zero= no pain and 10 = worest pain

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Asyut, Egypt

REFERENCES:
- [Background] Manyande A, Cyna AM, Yip P, Chooi C, Middleton P. Non-pharmacological interventions for assisting the induction of anaesthesia in children. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD006447. doi: 10.1002/14651858.CD006447.pub3. PMID 26171895
- [Background] Suresh S, Schaldenbrand K, Wallis B, De Oliveira GS Jr. Regional anaesthesia to improve pain outcomes in paediatric surgical patients: a qualitative systematic review of randomized controlled trials. Br J Anaesth. 2014 Sep;113(3):375-90. doi: 10.1093/bja/aeu156. Epub 2014 Jun 6. PMID 24907283
- [Background] De Jose Maria B, Banus E, Navarro Egea M, Serrano S, Perello M, Mabrok M. Ultrasound-guided supraclavicular vs infraclavicular brachial plexus blocks in children. Paediatr Anaesth. 2008 Sep;18(9):838-44. doi: 10.1111/j.1460-9592.2008.02644.x. Epub 2008 Jun 9. PMID 18544144
- [Derived] Elsawy S, Fathy E, Elbadawy A, Elnaggar A, Abdelatif AF, Elmorabaa H, Hamed R. Ultrasound-guided supraclavicular brachial plexus block as an additive to sevoflurane anesthesia in pediatrics undergoing brachiobasilic arteriovenous fistula operation: randomized controlled clinical trial. BMC Anesthesiol. 2025 May 16;25(1):248. doi: 10.1186/s12871-025-03091-1. PMID 40380096
- See also: Anaesthesia for children with renal disease. — https://doi.org/10.1093/bjaceaccp/mku064